CLINICAL TRIAL: NCT04877977
Title: Long-term Observation of Participants With Mood Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000375; 000375-M
Record Dates: First submitted 2021-05-06; First posted 2021-05-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11-25

CONDITIONS: Depression; Suicide Risk
Keywords: Depression; Suicide; Ketamine; Neuroimaging; Treatment Resistant Depression; Natural History
MeSH Terms: conditions — Depression; Suicide; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Individuals who previously signed consent for ETPB research as healthy volunteers
- Mood Disorder Patients: Individuals with mood disorders who previously signed consent for ETPB research

SUMMARY:
Background:

More than 12,000 people have taken part in research at the Experimental Therapeutics & Pathophysiology Branch at the National Institute of Mental Health Intramural Program. This has led to advances in the treatment of depression, bipolar disorder, and suicide risk. Researchers want to follow up with this group to see if they continue to have mental health symptoms and receive psychiatric treatments.

Objective:

To learn the long-term impact of depression, bipolar disorder, and suicide risk.

Eligibility:

Adults ages 18 and older who signed consent for Protocol 01-M-0254 over a year ago.

Design:

This study has 2 phases: an online phase and a telephone phase. It has no in-person or face-to-face contact.

In Phase 1, participants will fill out online surveys. They will access the surveys through the study website. The questions will focus on their current thoughts and feelings. The surveys will also ask about their current treatments for their mental health symptoms. At the end of the surveys, they will be asked if they would like to take part in Phase 2. If so, they will mark yes. Phase 2 includes a phone interview. They will be contacted by email to schedule the interview.

In Phase 2, participants will be asked more in-depth questions about how they are feeling. They will also be asked which psychiatric medicines and treatments they have used since they left NIH.

In both phases, participants can skip any questions they do not want to answer.

The online surveys will take 30 minutes to complete. The phone interview will last 1-4 hours.

The information that participants give in this study may be linked to their other NIH research records.

DETAILED DESCRIPTION:
Study Description: The proposal will leverage existing data on former participants with mood disorders collected in the Experimental Therapeutics and Pathophysiology Branch in order to identify predictors of long-term depressive symptoms, suicide attempts and ketamine utilization. The ETPB has collected a wealth of clinical, biologic, neuroimaging and sleep data on individuals with treatment resistant depression and bipolar disorder over the last 20 years. This study would re-contact these individuals for online and telephone assessment of current symptoms. We would then determine the ability of these clinical and biological measures to predict long-term outcomes. For individuals who do not participate in online or telephone data collection, we would like to identify incidence of premature death, including suicide, using linkage to data sources such as the National Death Index. We will also use this protocol for recruitment for in-person neurobiological studies and clinical trials of treatment resistant depression, bipolar disorder and suicide risk, both for ETPB and other branches of the NIMH IRP.

Objectives: The primary objective is to identify predictors of long-term treatment-resistant depression. The secondary and tertiary objectives are to identify predictors of long-term risk for suicide attempt and identify predictors of repeat use of ketamine, respectively

Endpoints:

Primary Endpoint: Score on Beck Depression Inventory

Secondary Endpoint: Self-reported suicide attempt after NIH study participation

Secondary Endpoint: Self-reported ketamine utilization after NIH study participation

Secondary Endpoint: Suicide death as reported by the National Death Index

Study Population: The sample size will be up to 1000 participants who previously signed consent into Protocol 01-M-0254: The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers and will include participants 18 years and older, any gender and health status.

Description of Sites/Facilities Enrolling Participants: The study will be conducted online through a secure study website. Data collection can also occur over the phone.

Study Duration: 1 year

Participant Duration: 20 minutes- 4 hours

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Participants who signed consent for Protocol 01-M-0254: The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers over a year ago.
2. Age 18 years or older
3. Able to provide informed consent online using study website or over the telephone
4. Able to read and write English

EXCLUSION CRITERIA:

None.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study involves re-contacting former participants of 01-M-0254: The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers for participation in this follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Score on Beck Depression Inventory (suicide item removed) | Follow-up assessment
  Rating of depression without assessment of suicidal ideation

SECONDARY OUTCOMES:
Ketamine utilization at non-NIH facility | Follow-up assessment
  Participants will report whether they accessed ketamine/esketamine after leaving NIH
Self-reported suicide attempt | Follow-up assessment
  Self-reported suicide attempt since leaving NIH
Identify predictors of death by suicide | Follow-up assessment
  Death as reported by the National Death Index (NDI)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth D Ballard, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical and demographic and biomarker participant data collected during the trial, after deidentification.
Supporting Information: SAP
Time Frame: Starting within 1 year of completion of the study
Access Criteria: Branch Chief will review requests and access will need to be approved by the NIMH/DIRP SD and OCD NIMH and the NIH IIRB.

REFERENCES:
- [Background] Gilbert JR, Ballard ED, Galiano CS, Nugent AC, Zarate CA Jr. Magnetoencephalographic Correlates of Suicidal Ideation in Major Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Mar;5(3):354-363. doi: 10.1016/j.bpsc.2019.11.011. Epub 2019 Dec 3. PMID 31928949
- [Background] Ballard ED, Vande Voort JL, Bernert RA, Luckenbaugh DA, Richards EM, Niciu MJ, Furey ML, Duncan WC Jr, Zarate CA Jr. Nocturnal Wakefulness Is Associated With Next-Day Suicidal Ideation in Major Depressive Disorder and Bipolar Disorder. J Clin Psychiatry. 2016 Jun;77(6):825-31. doi: 10.4088/JCP.15m09943. PMID 27337418
- [Background] Nugent AC, Ballard ED, Gould TD, Park LT, Moaddel R, Brutsche NE, Zarate CA Jr. Ketamine has distinct electrophysiological and behavioral effects in depressed and healthy subjects. Mol Psychiatry. 2019 Jul;24(7):1040-1052. doi: 10.1038/s41380-018-0028-2. Epub 2018 Feb 27. PMID 29487402
- [Derived] Hurst KT, Vogeley A, Greenstein DK, Durland L, Makel S, Wang PR, Yavi M, Zarate CA Jr, Ballard ED. Long-term follow-up of participants in ketamine clinical trials for mood disorders. J Affect Disord. 2024 Jul 15;357:134-137. doi: 10.1016/j.jad.2024.04.062. Epub 2024 Apr 22. PMID 38653350